CLINICAL TRIAL: NCT07133997
Title: A Phase 1/1b Study Evaluating Asparaginase Erwinia Chrysanthemi- Recombinant-Rywn (Recombinant Erwinia Asparaginase) and Venetoclax in Combination With Blinatumomab in Adults With Relapsed or Refractory B-Cell Acute Lymphoblastic Leukemia
Brief Title: Recombinant Erwinia Asparaginase and Venetoclax in Combination With Blinatumomab for the Treatment of Relapsed or Refractory CD19 Positive B-cell Acute Lymphoblastic Leukemia
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24738; NCI-2025-05656 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24738 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2025-08-14; First posted 2025-08-21 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Recurrent B Acute Lymphoblastic Leukemia; Refractory B Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Burkitt Lymphoma | interventions — asparaginase erwinia chrysanthemi recombinant; Asparaginase; Specimen Handling; blinatumomab; N,N-dicyclohexyl-isoborneol-10-sulfonamide; Biopsy; Cyclophosphamide; Spinal Puncture; venetoclax; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (asparaginase, venetoclax, blinatumomab) (Experimental): PRE-PHASE TREATMENT/BRIDGE THERAPY: Starting days -7 to -5, patients may optionally receive cyclophosphamide and vincristine on day 1 and prednisone on days 1-5.
  TREATMENT: Patients receive asparaginase Erwinia chrysanthemi IM on days 1,3, 5, 7, 9, 11, and 13, venetoclax PO QD on days 1-14 or QOD on days 1, 3, 5, 7, 9, 11, and 13 of each cycle and blinatumomab CIV on days 8-35 of cycle 1 and on days 1-28 of cycle 2. Cycles repeat every 49 days for cycle 1 and 42 days for cycle 2 for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo ECHO and MUGA at screening and bone marrow aspiration and biopsy, blood sample collection, and lumbar puncture throughout the study.
  Interventions: Drug: Asparaginase Erwinia chrysanthemi; Procedure: Biospecimen Collection; Biological: Blinatumomab; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Cyclophosphamide; Procedure: Echocardiography Test; Procedure: Lumbar Puncture; Procedure: Multigated Acquisition Scan; Drug: Venetoclax; Drug: Vincristine

INTERVENTIONS:
Drug: Asparaginase Erwinia chrysanthemi — Given IM
  Other Names: Asparaginase Erwinia chrysanthemi (Recombinant)-rywn; Asparaginase Erwinia chrysanthemi, Recombinant-rywn; Asparaginase Erwinia chrysanthemi-rywn; Crisantaspase; Crisantaspase Biobetter JZP-458; Crisantaspasum; Enrylaze; Erwinase; Erwinaze; JZP 458; JZP-458; JZP458; PF743; RC-P JZP-458; Recombinant Asparaginase erwinia chrysanthemi JZP-458; Recombinant Crisantaspase JZP-458; Recombinant Erwinia asparaginase JZP-458; Rylaze
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Biological: Blinatumomab — Given CIV
  Other Names: AMG 103; AMG-103; AMG103; Anti-CD19 x Anti-CD3 Bispecific Monoclonal Antibody; Anti-CD19/Anti-CD3 Recombinant Bispecific Monoclonal Antibody MT103; Blincyto; MEDI 538; MEDI-538; MEDI538; MT 103; MT-103; MT103
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration and biopsy
Procedure: Bone Marrow Biopsy — Undergo bone marrow aspiration and biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Drug: Cyclophosphamide — Given cyclophosphamide
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Procedure: Lumbar Puncture — Undergo lumbar puncture
  Other Names: LP; Spinal Tap
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Drug: Venetoclax — Given PO
  Other Names: ABT 199; ABT-0199; ABT-199; ABT199; GDC 0199; GDC-0199; GDC0199; RG7601; Venclexta; Venclyxto
Drug: Vincristine — Given vincristine
  Other Names: LCR; Leurocristine; VCR; Vincrystine

SUMMARY:
This phase I/Ib trial tests the safety and side effects of asparaginase Erwinia chrysanthemi-recombinant-rywn (recombinant Erwinia asparaginase) and venetoclax in combination with blinatumomab and how well the combination works in treating patients with CD19 positive B-cell acute lymphoblastic leukemia (ALL) that has come back after a period of improvement (relapsed) or that has not responded to previous treatment (refractory). Asparaginase Erwinia chrysanthemi, a type of protein synthesis inhibitor, is a drug that is made up of the enzyme asparaginase, which comes from the bacterium Erwinia chrysanthemi. It is used in people who cannot take asparaginase that comes from the bacterium E. coli. Asparaginase Erwinia chrysanthemi breaks down the amino acid asparagine and may stop the growth of cancer cells that need asparagine to grow. It may also kill cancer cells. Venetoclax is in a class of medications called B-cell lymphoma-2 (BCL-2) inhibitors. It may stop the growth of cancer cells by blocking Bcl-2, a protein needed for cancer cell survival. Blinatumomab is a drug used to treat certain types of B-cell acute lymphoblastic leukemia that are CD19 positive (expresses the protein CD19). Blinatumomab binds to CD19, which is found on most B cells (a type of white blood cell) and some types of leukemia cells. It also binds to a protein called CD3, which is found on T cells (another type of white blood cell). This may help the immune system kill cancer cells. Blinatumomab is a type of bispecific T-cell engager. Giving asparaginase Erwinia chrysanthemi and venetoclax in combination with blinatumomab may be safe, tolerable, and/or effective in treating patients with relapsed or refractory ALL.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the safety and tolerability of asparaginase Erwinia chrysanthemi- recombinant-rywn (recombinant Erwinia asparaginase) and venetoclax in combination with blinatumomab for the target population by evaluation of toxicities including: type, frequency, severity, attribution, time course and duration. (Phase I) II. Determine the recommended phase 2 schedule (RP2S) of recombinant Erwinia asparaginase and venetoclax in combination with blinatumomab. (Phase I) III. Estimate the anti-tumor efficacy of recombinant Erwinia asparaginase and venetoclax in combination with blinatumomab as assessed by composite remission (including complete remission (CR), CR with partial hematologic recovery (CRh) and CR with incomplete hematologic recover (CRi) rate. (Expansion Phase)

SECONDARY OBJECTIVES:

I. Evaluate the safety of recombinant Erwinia asparaginase in combination with blinatumomab and venetoclax at expansion phase.

II. Estimate minimal residual disease (MRD) negativity (-) rate at the end of each cycle (by flow MRD and Clonoseq).

III. Among transplant eligible patients, determine the number and proportion of patients who bridge directly from trial therapy to allogeneic hematopoietic stem cell transplant (alloHSCT).

EXPLORATORY OBJECTIVES:

I. Explore BH3 profiling on pretreatment bone marrow aspirate to predict response to blinatumomab with recombinant Erwinia asparaginase and venetoclax.

II. Explore role of somatic mutations in pretreatment bone marrow biopsy to predict response to blinatumomab with recombinant Erwinia asparaginase and venetoclax.

III. Examine changes in cell composition-both leukemic and non-leukemic-before and after treatment.

IV. Estimate the proportion of patients maintaining adequate nadir serum asparaginase activity (≥ 0.1 IU/mL) at 48 hours post last dose of recombinant Erwinia asparaginase.

V. Immune profiling of ALL blasts.

OUTLINE:

PRE-PHASE TREATMENT/BRIDGE THERAPY: Starting days -7 to -5, patients may optionally receive cyclophosphamide and vincristine on day 1 and prednisone on days 1-5.

TREATMENT: Patients receive asparaginase Erwinia chrysanthemi intramuscularly (IM) on days 1,3, 5, 7, 9, 11, and 13, venetoclax orally (PO) once daily (QD) on days 1-14 or once every other day (QOD) on days 1, 3, 5, 7, 9, 11, and 13 of each cycle and blinatumomab continuous intravenously (CIV) on days 8-35 of cycle 1 and on days 1-28 of cycle 2. Cycles repeat every 49 days for cycle 1 and 42 days for cycle 2 for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo echocardiography (ECHO) and multigated acquisition scan (MUGA) at screening and bone marrow aspiration and biopsy, blood sample collection, and lumbar puncture throughout the study.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative
* Age between 12 and 55
* Eastern Cooperative Oncology Group (ECOG) ≤ 2 or Karnofsky performance status (KPS) ≥ 70
* Patients with relapsed or refractory (R/R) CD19 positive (+) B-cell acute lymphoblastic leukemia (B-ALL) according to World Health Organization (WHO) criteria

  * Greater than or equal to 5% blasts in the bone marrow
* White blood cell count less than 25 x 10^9/L prior to initiation of venetoclax. (within 14 days prior to day 1 of protocol therapy) Cytoreduction with hydroxyurea, steroid or a single dose of cyclophosphamide chemotherapy prior to treatment may be required
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN) (within 14 days prior to day 1 of protocol therapy) (unless has Gilbert's disease or underlying leukemia, ≤ 3 x ULN)
* Prothrombin time (PT) ≤ 1.5 ULN (within 14 days prior to day 1 of protocol therapy)
* Partial thromboplastin time (PTT) ≤ 1.5 ULN (within 14 days prior to day 1 of protocol therapy)
* Aspartate aminotransferase (AST) ≤ 2.5 x ULN (within 14 days prior to day 1 of protocol therapy) (Unless it is related to underlying leukemia, then AST ≤ 5 x ULN)
* Alanine aminotransferase (ALT) ≤ 2.5 x ULN (within 14 days prior to day 1 of protocol therapy) (Unless it is related to underlying leukemia, then ALT ≤ 5 x ULN)
* Creatinine clearance of ≥ 60 mL/min per 24 hour urine test or the Cockcroft-Gault formula (within 14 days prior to day 1 of protocol therapy)
* Left ventricular ejection fraction (LVEF) ≥ 50% (within 14 days prior to day 1 of protocol therapy)

  * Note: Echocardiogram to be performed within 42 days prior to day 1 of protocol therapy
* Women of childbearing potential (WOCBP): Negative urine or serum pregnancy test (within 14 days prior to day 1 of protocol therapy)

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 3 months after the last dose of protocol therapy

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only).

Exclusion Criteria:

* Allogeneic hematopoietic cell transplantation (HCT) within 8 weeks prior to the start of protocol-specific therapy. Subjects must be off all immunosuppression for ≥ 2 weeks
* Cancer chemotherapy within 2 weeks before the start of protocol-specified therapy with the exception of: intrathecal chemotherapy and/or low-dose maintenance therapy (e.g. vina alkaloids, mercaptopurine, methotrexate, or hydroxyurea etc)
* Strong and moderate CYP3A4 inducers and strong CYP3A inhibitors within 7 days prior to day 1 of protocol therapy
* Foods/supplements that are strong inhibitors or strong or moderate inducers of CYP3A (such as grapefruit, Seville oranges, starfruit and St. John's wort) within 3 days prior to initiation of and during study treatment
* Immunotherapy (e.g. rituximab) within 4 weeks before the start of protocol-specified therapy. Prior failed CD19-directed therapy such as prior blinatumomab or CD19-directed chimeric antigen receptor (CAR)-T cells will be allowed if treatment ended > 4 weeks prior to start of protocol-specific therapy and there is demonstrated continued CD19+ expression
* Must not have received or planning to receive live vaccine while being on study or 2 weeks before and after completion of treatment
* Patients with any prior intolerance leading to discontinuation of pegylated (PEG)-asparaginase due to grade 3 or more pancreatitis or central nervous system thrombosis requiring anticoagulant treatment attributed to the PEG-asparaginase
* Active ALL in the central nervous system (CNS): Presence of > 5 white blood cells (WBC) per cubic millimeter in the cerebrospinal fluid (CSF) with lymphoblasts present (confirmed by CSF analysis) and/or clinical signs of CNS leukemia. If CSF leukemia is present, subjects will need to receive intrathecal chemotherapy and have documented negative CSF prior to enrollment
* Active acute or chronic graft versus host disease requiring systemic treatment with immunosuppressive medication
* History of intracranial thrombosis or history of recurrent thrombosis or grade 3 and greater pulmonary embolism (except for catheter-related thrombosis)
* Participants with history of grade ≥ 3 pancreatitis
* History of alcohol overuse if deemed relevant in investigator's opinion
* Known hypersensitivity to blinatumomab/ recombinant Erwinia asparaginase or to any component of the product formulation, otherwise prior treatment with single agent blinatumomab is allowed
* Uncontrolled active infection
* Clinically significant uncontrolled illness or cirrhosis
* Other active malignancy (except superficial skin cancers squamous cell carcinoma [SCC]/basal cell carcinoma [BCC], early-stage malignancies ductal carcinoma in-situ [DCIS] status post [s/p] excision or elevated prostate specific antigen [PSA])
* Females only: Pregnant or breastfeeding
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Ages: 12 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Estimated)
Dates: Start 2026-01-26 (Estimated); Primary Completion 2027-05-08 (Estimated); Study Completion 2027-05-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) (Phase I) | Up to 30 days after last dose of study treatment
  Will be graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0. Will be summarized in terms of type (organ affected or laboratory determination), severity, attribution, time of onset, duration, probable association with the study treatment and reversibility or outcome by counts/ rates and 95% Clopper Pearson confidence interval (CI).
Dose-limiting toxicities (DLT) (Phase I) | From the start of therapy (day 1) through the end of the first cycle (day 49)
  Will be graded according to NCI CTCAE v 5.0. Will be summarized in terms of type (organ affected or laboratory determination), severity, attribution, time of onset, duration, probable association with the study treatment and reversibility or outcome by counts/ rates and 95% Clopper Pearson CI.
Maximum tolerated schedule (Phase I) | During cycle 1 (cycle length = 49 days)
  Will be based on the assessment of DLT during cycle 1.
Recommended phase 2 schedule (Phase 1) | After cycle 1 (cycle length = 49 days)
  Will be selected based on maximum tolerated schedule and a review of cumulative toxicity and tolerability data after cycle 1 and may be lower than the maximum tolerated schedule.
Best response (Expansion Phase) | Up to 30 days after last dose of study treatment
  The 95% Clopper Pearson binomial CI will be calculated.

SECONDARY OUTCOMES:
Composite remission rate | At end of cycle 1 (cycle length = 49 days)
  The complete remission (CR)/CR with incomplete recovery/CR with partial hematologic recovery and 95% Clopper Pearson binomial CI will be calculated.
Minimal residual disease negativity | At the end of each cycle (cycle 1 length = 49 days, cycle 2 length = 42 days)
  Will be defined as residual leukemia < 0.01% by flow cytometry or Clonoseq in bone marrow biopsy. Clopper Pearson binomial CI will be calculated.
Incidence of adverse events (Expansion Phase) | Up to 30 days after last dose of study treatment
  Will be graded according to NCI CTCAE v 5.0. Will be summarized in terms of type (organ affected or laboratory determination), severity, attribution, time of onset, duration, probable association with the study treatment and reversibility or outcome by counts/ rates and 95% Clopper Pearson CI.
Patients who bridge to transplant directly from the trial therapy | Up to 30 days after last dose of study treatment
  The Clopper Pearson binomial CI will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Amandeep Salhotra, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States